CLINICAL TRIAL: NCT01524367
Title: Effect of Single-dose Dexmedetomidine on Emergence Excitement in Adults With Nasotracheal Intubation After Orthognathic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yon Hee Shim, MD, PhD, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2011-0200
Record Dates: First submitted 2011-10-28; First posted 2012-02-02 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Sodium Chloride; Saline Solution; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline group (Placebo Comparator): We administrate the saline single bolus (0.01ml/kg,intravenously) at time of oral cavity sealing.
  Interventions: Drug: saline
- dexmedetomidine group (Experimental): We administrate the dexmedetomidine single bolus (1ug/kg, intravenously) at time of oral cavity sealing.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: saline — We administrate the normal saline (single bolus, 0.01ml/kg) intravenously at time of oral cavity sealing.
  Other Names: normal saline
  Arms: saline group
Drug: Dexmedetomidine — We administrate the dexmedetomidine (single bolus, 1 ug/ks) intravenously at time of oral cavity sealing.
  Other Names: Precedex
  Arms: dexmedetomidine group

SUMMARY:
Excitement during the emergence from general anesthesia is a great post-operative problem. It may lead to serious consequences for the patient, such as injury, increased pain, hemorrhage, self-extubation, and removal of catheters, and it can necessitate physically or chemically restraining the patient. It has been reported that the incidence of postoperative emergence excitement in adults after general anesthesia is 21.3% occurrence.

Many things are mentioned as risk factors for emergence excitement. Among them, excitement after orthognathic surgery (two-jaw) was more common than after other types of surgery. The patients undergoing emergence with nasotracheal intubation after orthognathic surgery may have a sense of suffocation during emergence from anesthesia, which may increase the incidence of emergence excitement.

Pain is also a main cause of postoperative excitement. Dexmedetomidine, which is an S-enantiomer of medetomidine with high specificity for α2-adrenoceptor (α2 : α1, 1620 : 1) compared to clonidine (a2 : a1, 220 : 1), is approved as a sedative and co-analgesic drug.

To the best of the investigators knowledge, effect of dexmedetomidine on emergence excitement was investigated only in children.

The investigators hypothesized that single dose of dexmedetomidine would reduce the incidence and the severity of the emergence excitement in adults with nasotracheal intubation after orthognathic surgery (two-jaw).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 or 2 patients
* patients scheduled for orthognathic surgery (two-jaw)

Exclusion Criteria:

* severe cardiovascular disease
* allergy to dexmedetomidine
* psychological disease
* patients who cannot understand Korean

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
severity of emergence excitement based on Richmond agitation-sedation scale | Patients will be followed for the duration of stay in operation room and post anesthetic recovery room, an expected average of 2 hours.
  The severity of emergence excitement will be measured up to 10 minutes after extubation based on Richmond agitation-sedation(time of eye opening on command, time of leaving the operation room, 5 minutes after arriving post anesthetic recovery room, 10 minutes after extubation).

SECONDARY OUTCOMES:
emergence time | up to the time of eye opening,an expected average of 30 minutes.
  The emergence time will be recorded as the time from desflurane discontinue to eye opening on command.
coughing grade | up to the time of leaving the postanesthetic recovery room,an expected average of 2 hours.
  The coughing grade will be measured up to the time of leaving the postanesthetic recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: Yonhee Shim, Study Director — Yonsei University
Locations (1):
- Gangnam severance hospital, Seoul, South Korea